CLINICAL TRIAL: NCT04683549
Title: HPV Serum Level and FDG PET CT in Patients With Cervical Cancer Treated With Radical Radiochemotherapy (HPV-RICCO - HPV Relation in Cervical Cancer Outcomes)
Brief Title: HPV Serum Level and FDG PET CT in Patients With Cervical Cancer Treated With Radical Radiochemotherapy
Acronym: HPV-RICCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/06/2020/E/WCO/007
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Cervical Cancer
Keywords: locally advanced cervical cancer; HPV; radiochemotherapy; FDG PET CT
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Locally advanced non-operable newly diagnosed FIGO stage IB-IVA cervical cancer patients planned for definitive radiochemotherapy will be accrued to study and will have:
  1. FDG PET Scan before treatment and 3 months after treatment
  2. Pre- treatment DNA from the neoplastic time preserved in the form of paraffin blocks to determine HPV status
  3. Blood sample to measure HPV DNA at time point baseline (before treatment), in the middle of treatment and at the end of definitive radiochemotherapy,
  4. [F-18] - FDG PET scan before treatment and 3 months post completion of radiochemotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One-Arm HPV serum level and FDG PET CT (Other): HPV serum level and FDG PET CT in patients with cervical cancer treated with radical radiochemotherapy
  Interventions: Diagnostic Test: HPV serum level and FDG PET CT in patients with cervical cancer treated with radical radiochemotherapy

INTERVENTIONS:
Diagnostic Test: HPV serum level and FDG PET CT in patients with cervical cancer treated with radical radiochemotherapy — Locally advanced non-operable newly diagnosed FIGO stage IB-IVA cervical cancer patients planned for definitive radiochemotherapy will be accrued to study and will have:
  1. FDG PET Scan before treatment and 3 months after treatment
  2. Pre- treatment DNA from the neoplastic time preserved in the form of paraffin blocks to determine HPV status
  3. Blood sample to measure HPV DNA at time point baseline (before treatment), in the middle of treatment and at the end of definitive radiochemotherapy,
  4. [F-18] - FDG PET scan before treatment and 3 months post completion of radiochemotherapy.

SUMMARY:
The main purpose of the study is to describe changes in plasma HPV DNA levels in patients with locally advanced cervical cancer during radical radiochemotherapy (CRT) and to correlate changes with response to treatment. Monitoring of the response to treatment will also be assessed in FDG PET CT imaging.

DETAILED DESCRIPTION:
Ninety-five per cent of cervical cancer cases are caused by persistent infections with carcinogenic HPVs. Locally advanced stage IB2 to IVA cervical cancers are treated with definitive chemoradiation therapy (CRT). Despite known clinical prognostic factors of poor treatment outcome such as advanced stage and positive nodal status, we still don't know predictors of relapse.

HPV status will be assessed in the neoplastic tissue and DNA from the blood serum of patients with cervical cancer will be isolated and analyzed by real-time PCR. Plasma HPV DNA would identify patients with residual disease after CRT due to persistent detectable HPV. This would earlier detect high risk patients who would benefit from adjuvant therapy.

While metabolic response in post - therapy FDG PET CT is predictive of survival, there is usually 3 months waiting period time needed to perform this imaging. This pilot study will provide preliminary estimates of the correlation between plasma HPV DNA level, PET finding and clinical outcome in polish cervical cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Age Limits: more than 18Y Histologically confirmed squamous cell carcinoma, FIGO stage IB-IVA planned for radical radiochemotherapy Eastern Cooperative Oncology Group (ECOG) performance status 0,1,2

Exclusion Criteria:

Patients who have received any anticancer treatment for their cervical cancer. Eastern Cooperative Oncology Group (ECOG) performance status > 2 Other cervical cancer tumor histologies (e.g. small cell, serous) Contraindications to 18FDG PET-CT Contraindication to radiochemotherapy Known pregnancy or lactating

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
local control | 18 months
Response to treatment | 6 months

SECONDARY OUTCOMES:
Progression-free survival | 18 months
Plasma HPV DNA levels | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Burchardt, PhD, MD, Principal Investigator — Oncological Gynecology Clinic / GPCC
Locations (1):
- Greater Poland Cancer Centre / Oncological Gynecology Clinic, Poznan, Greater Poland Voivodeship, Poland